CLINICAL TRIAL: NCT05422755
Title: A Prospective, Open Label, Single Arm, and Multicenter Study to Evaluate Immunogenicity of Epodion in Anemia Associated With Chronic Kidney Disease (CKD) Patients
Brief Title: The Clinical Study to Evaluate Immunogenicity of Epodion® in Anemia Associated With CKD Patients
Status: Completed | Type: Observational
Sponsor: PT. Daewoong Infion (Industry)
Collaborators: Equilab International (Unknown)
Responsible Party: Sponsor
Other Study IDs: DW_EPOC01
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: rh-EPO; Chronic Kidney Disease; Erythropoietin alpha
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples With DNA — Blood samples on weeks 0, 24, and 52.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: Experimental: Test Drug Recombinant Human Erythropoietin Alfa

SUMMARY:
The study was conducted to assess safety and immunogenicity of recombinant human erythropoietin (rhEPO) manufactured by Daewoong Pharmaceutical Co., Ltd was similar to biological products approved by the drug safety regulatory authority.

DETAILED DESCRIPTION:
This study consisted of a screening period (4 weeks) and treatment period (52 weeks). Evaluation for immunogenicity effect using ADA (Anti Drug Antibody) detection will be done at weeks 0, 24, and 52 and blood sampling for Routine Hematological tests as supporting data will be conducted every month following hospital regulation. For each subject, the end of the study is the last day of the Blood sample will be drawn In the case of a subject that has left the study (withdrawn), the exit date will be the end of the study. The safety evaluation was conducted based on the incidence of the adverse events local and systemic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have anemia associated with Chronic Kidney Disease (CKD) under hemodialysis treatment.
* Male or female patients aged ≥18 years.
* Patients with mean Hb concentration when screening is around ≤10 g/dL.
* Patients on stable, adequate dialysis for at least three months (defined as no clinically relevant changes of hemodialysis regimen and/or 23/42 ©EMEA 2007 dialyzer).
* Has ever been using Epodion treatment in the at least last 1 month.
* Haemodialysis patients who likely to remain on Epodion treatment for 52 weeks.
* Informed consent given in a written form after being provided with detailed information about the nature, risks, and scope of the clinical trial as well as the expected desirable and adverse effects of the drug.

Exclusion Criteria:

* History of Pure Red Cell Aplasia (PRCA) or anti-epoetin antibodies.
* Contraindications for ESA therapy.
* Systemic immunosuppressive medication or any other drugs known to adversely affect the hemoglobin level.
* History of uncontrolled hypertension (defined as systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg during screening).
* Any blood transfusion within the last 2 weeks prior to screening period.
* Major surgery within 3 months prior to screening period.
* Myelodysplastic syndrome.
* History bleeding disorders (e.g. Hemophilia, Von Willebrand, and any conditions that result when the blood cannot clot properly).
* Known bone marrow fibrosis (osteitis fibrosa cystica).
* Known epilepsy.
* Liver cirrhosis with clinical evidence of complications (portal hypertension, splenomegaly, ascites).
* Systemic lupus erythematosus.
* Previously diagnosed with HIV or acute hepatitis infection.
* History of malignancy of any organ system within the last 5 year.
* Pregnancy or lactation period in female patients.
* Heavy smoker (who smoke over 20 cigarettes daily in average).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted on Patients who have anemia associated with Chronic Kidney Disease (CKD) under hemodialysis treatment and Have been using Epodion treatment for at least the last 1 month in several hospitals in Jakarta.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Anti-Erythropoietin Antibodies (ADA) formation at week 52nd | week 52
  to evaluate if there is any incidence of ADA formation on the blood sample
Neutralizing Antibodies detection (Nab) (will be assessed if ADA is positive). | week 52
  to evaluate the neutralizing effect of the detected ADA using cell-based assay method to confirm the impact of the antibody to pharmacological activity.

SECONDARY OUTCOMES:
Any Adverse Event | 52 weeks
  to evaluate any adverse event related to the test product during study
Incidence of Anti-Erythropoietin Antibodies (ADA) formation at week 24th | week 24
  to evaluate if there is any incidence of ADA formation on the blood sample
Comparison on the incidence of Anti-Erythropoietin Antibodies (ADA) formation at week 24th and week 52nd. | week 24 and 52
  to evaluate the neutralizing effect of the detected ADA using cell-based assay method to confirm the impact of the antibody to pharmacological activity.

CONTACTS AND LOCATIONS:
Overall Officials: Nova Angginy, Study Director — PT. Daewoong Infion
Locations (1):
- Gatot Soebroto Army Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No